CLINICAL TRIAL: NCT02210728
Title: Efficacy of Cognitive Behavioral Therapy in Treatment of Adults With Attention Deficit Hyperactivity Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lily Hechtman (Other)
Responsible Party: Sponsor-Investigator, Lily Hechtman, Professor of Psychiatry and Pediatrics; Director of Research - Division of Child Psychiatry, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PED-06-002
Record Dates: First submitted 2014-07-31; First posted 2014-08-07 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: cognitive behavioral therapy; stimulant medication; efficacy; symptoms; functional outcomes
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Dextroamphetamine; SLI381; Lisdexamfetamine Dimesylate; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Medication only (Active Comparator): Stimulant medication (methylphenidate or amphetamine product approved for clinical use in Canada), with dose optimized for each patient based on report of efficacy and side effects.
  Interventions: Drug: methylphenidate or amphetamine product
- Cognitive behavioral therapy + medication (Active Comparator): Patients are first titrated to an optimal dose of stimulant medication. They then undergo the 12 weeks of group cognitive behavioral therapy.
  Interventions: Drug: methylphenidate or amphetamine product; Behavioral: Cognitive behavioral therapy
- Cognitive behavioral therapy alone (Experimental): 12 weeks of structured group cognitive behavioral therapy, focusing on acquisition of skills in organization, time management, goal attainment, cognitive restructuring, stress management, anger management, impulse control, self-esteem, and relationship management.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Drug: methylphenidate or amphetamine product — Medication is titrated over a 4-week period with stepwise increments each week. Patients and significant others complete ADHD symptom scales at baseline and before each medication visit. Patients also complete side effects scales at baseline and before each medication visit. The gradual increase will continue until there is no further improvement in symptoms and in the Clinical Global Improvement Scale or side effects are such that further increases are not indicated. Once the optimal dose is reached, the subjects remain on this dose for the remainder of the study.
  Other Names: Ritalin; Concerta; Biphentin; Dexedrine; Adderall XR; Vyvanse
  Arms: Cognitive behavioral therapy + medication; Medication only
Behavioral: Cognitive behavioral therapy — 12 sessions of group cognitive behavioral therapy. Participants also receive individual coaching 3 times a week (twice over telephone and once in person). Coaching sessions are 15 minutes each in duration and are aimed at implementation, practice, and generalization of skills acquired in therapy.
  Arms: Cognitive behavioral therapy + medication; Cognitive behavioral therapy alone

SUMMARY:
The purpose of the project is to evaluate the efficacy of cognitive behavioral therapy (CBT) for adults with attention deficit hyperactivity disorder (ADHD) with and without stimulant medication and compare it to medication alone. Subjects will be randomly assigned to stimulant medication only, CBT only and combined CBT and stimulant medication group. Patients will be evaluated at baseline, following mediation optimization (for medicated groups), following 12 months of treatment, after 3 months of follow up, and after 6 months of follow up. The investigators hypothesize that the combined group will have the best outcome at all evaluation points. ADHD in adults is associated with significant morbidity and impaired academic, occupational, social, and emotional functioning. Developing optimal treatment approaches for this population is key in improving their functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision (DSM-IV-TR) criteria for adult ADHD of any of three subtypes via Conners' Adult ADHD Diagnostic Interview for the DSM-IV (CAAR-D) and clinician's assessment;
* Barkley Childhood and Current Symptom of ADHD (1998) completed by self and informants (parents or siblings). Required cut off's on these scales are scores 1.5 Standard Deviation above relevant gender and age norms;
* Conners' Adult ADHD Rating Scale (1999). Required cut off's on these scales are scores 1.5 Standard Deviation above relevant gender and age norms;
* Between 18 and 60 years old
* Be able to give informed consent and comply with study procedures;
* I.Q. of 80 or above on Wechsler Adult Intelligence Scale, 3rd edition (WAIS-III) subtests of three verbal and three nonverbal subtests
* Adequate command of English to be able to participate in CBT group.

Exclusion Criteria:

* Psychotic symptoms, past or current
* Current psychiatric comorbidity, e.g. bipolar disorder, depression, suicidality, current substance use disorder (must be free of substance abuse for 6 months)
* Medical condition that preclude use of the stimulant medication, e.g. hypertension, cardiac disease, Tourette's Syndrome, etc.
* Organic mental disorders or other significant neurological disorders, e.g. epilepsy, head injury, chorea, multiple sclerosis, deafness, blindness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-04; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Self-reported ADHD symptoms (measured via Barkley's Current ADHD Symptoms Scale) - Change from baseline | At baseline
Self-reported ADHD symptoms (measured via Barkley's Current ADHD Symptoms Scale) | For patients in a medication or combined group - after medication has been optimally titrated, approximately 5 weeks.
Self-reported ADHD symptoms (measured via Barkley's Current ADHD Symptoms Scale) | After 12 weeks of Cognitive Behavioural Therapy
Self-reported ADHD symptoms (measured via Barkley's Current ADHD Symptoms Scale) | Three months after the end of Cognitive Behavioural Therapy
Self-reported ADHD symptoms (measured via Barkley's Current ADHD Symptoms Scale) | Six months after the end of Cognitive Behavioural Therapy

SECONDARY OUTCOMES:
Global psychological distress (measured via the Symptom Checklist 90) - Change from baseline | At baseline; once optimally titrated, takes approximately 5 weeks to reach this dose (for medicated participants); after cognitive behavioural therapy; 3 months of follow up; 6 months of follow up
Depression symptoms (via the Beck Depression Inventory) - Change from baseline | At baseline; once optimally titrated, takes approximately 5 weeks to reach this dose (for medicated participants); after cognitive behavioural therapy; 3 months of follow up; 6 months of follow up
Anxiety symptoms (measured via the Beck Anxiety Inventory) - Change from baseline | At baseline; once optimally titrated, approximately 5 weeks (for medicated participants); after cognitive behavioural therapy; 3 months of follow up; 6 months of follow up
Global functional impairment (measured via the Sheehan Disability Scale) - Change from baseline | At baseline; once optimally titrated, takes approximately 5 weeks to reach this dose (for medicated participants); after cognitive behavioural therapy; 3 months of follow up; 6 months of follow up
Dyadic adjustment (for those married or cohabiting, measured via the Dyadic Adjustment Scale) - Change from baseline | At baseline; once optimally titrated, takes approximately 5 weeks to reach this dose (for medicated participants); after cognitive behavioural therapy; 3 months of follow up; 6 months of follow up
Organizational skills (measured via the Organization and Activation for Work Scale) - Change from baseline | At baseline; once optimally titrated, takes approximately 5 weeks to reach this dose (for medicated participants); after cognitive behavioural therapy; 3 months of follow up; 6 months of follow up
Self-esteem (measured via the Index of Self-Esteem) - Change from baseline | At baseline; once optimally titrated, takes approximately 5 weeks to reach this dose (for medicated participants); after cognitive behavioural therapy; 3 months of follow up; 6 months of follow up
Anger Expression (measured via the State Trait Anger Expression Inventory - II) - Change from baseline | At baseline; once optimally titrated, takes approximately 5 weeks to reach this dose (for medicated participants); after cognitive behavioural therapy; 3 months of follow up; 6 months of follow up
Observer-Rated ADHD symptoms (measured via the Barkley's Current ADHD Symptoms Scale -- observer version) - Change from baseline | At baseline; once optimally titrated, takes approximately 5 weeks to reach this dose (for medicated participants); after cognitive behavioural therapy; 3 months of follow up; 6 months of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hechtman, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Kessler RC, Adler L, Barkley R, Biederman J, Conners CK, Demler O, Faraone SV, Greenhill LL, Howes MJ, Secnik K, Spencer T, Ustun TB, Walters EE, Zaslavsky AM. The prevalence and correlates of adult ADHD in the United States: results from the National Comorbidity Survey Replication. Am J Psychiatry. 2006 Apr;163(4):716-23. doi: 10.1176/ajp.2006.163.4.716. PMID 16585449
- [Background] Safren SA. Cognitive-behavioral approaches to ADHD treatment in adulthood. J Clin Psychiatry. 2006;67 Suppl 8:46-50. PMID 16961430
- [Background] Wilens TE, Spencer TJ, Biederman J. A review of the pharmacotherapy of adults with attention-deficit/hyperactivity disorder. J Atten Disord. 2002 Mar;5(4):189-202. doi: 10.1177/108705470100500401. PMID 11967475
- [Background] Bramham J, Young S, Bickerdike A, Spain D, McCartan D, Xenitidis K. Evaluation of group cognitive behavioral therapy for adults with ADHD. J Atten Disord. 2009 Mar;12(5):434-41. doi: 10.1177/1087054708314596. Epub 2008 Feb 29. PMID 18310557
- [Background] Gualtieri CT, Ondrusek MG, Finley C. Attention deficit disorders in adults. Clin Neuropharmacol. 1985;8(4):343-56. doi: 10.1097/00002826-198512000-00005. PMID 4075304
- [Background] Knouse LE, Cooper-Vince C, Sprich S, Safren SA. Recent developments in the psychosocial treatment of adult ADHD. Expert Rev Neurother. 2008 Oct;8(10):1537-48. doi: 10.1586/14737175.8.10.1537. PMID 18928346
- [Background] Mattes JA, Boswell L, Oliver H. Methylphenidate effects on symptoms of attention deficit disorder in adults. Arch Gen Psychiatry. 1984 Nov;41(11):1059-63. doi: 10.1001/archpsyc.1983.01790220049008. PMID 6388523
- [Background] Safren SA, Sprich S, Mimiaga MJ, Surman C, Knouse L, Groves M, Otto MW. Cognitive behavioral therapy vs relaxation with educational support for medication-treated adults with ADHD and persistent symptoms: a randomized controlled trial. JAMA. 2010 Aug 25;304(8):875-80. doi: 10.1001/jama.2010.1192. PMID 20736471
- [Background] Solanto MV, Marks DJ, Wasserstein J, Mitchell K, Abikoff H, Alvir JM, Kofman MD. Efficacy of meta-cognitive therapy for adult ADHD. Am J Psychiatry. 2010 Aug;167(8):958-68. doi: 10.1176/appi.ajp.2009.09081123. Epub 2010 Mar 15. PMID 20231319
- [Background] Spencer T, Biederman J, Wilens T, Doyle R, Surman C, Prince J, Mick E, Aleardi M, Herzig K, Faraone S. A large, double-blind, randomized clinical trial of methylphenidate in the treatment of adults with attention-deficit/hyperactivity disorder. Biol Psychiatry. 2005 Mar 1;57(5):456-63. doi: 10.1016/j.biopsych.2004.11.043. PMID 15737659
- [Background] Weiss, G., & Hechtman, L. (1993). Hyperactive children grown up : ADHD in children, adolescents, and adults (2nd ed.). New York: Guilford Press.
- [Background] Barkley, R. A., Murphy, K. R., & Firscher, M. (2008). ADHD in adults: What the Science Says. New York: Guilford Press
- [Result] Hechtman, L., Treatment of adults with adhd: Cbt only versus medication and cbt, in Third International Congress on ADHD - From Childhood to Adolescence. 2011: Berlin, Germany.